CLINICAL TRIAL: NCT05602272
Title: Respiratory and Hemodynamic Implications of Endoscopic Myotomy of the Esophagus and Stomach (POEM/GPOEM)
Brief Title: Respiratory and Hemodynamic Implications of Endoscopic Myotomy of the Esophagus and Stomach
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Chollet-Rivier, Chief physician of anesthesiology department, Centre Hospitalier Universitaire Vaudois
Other Study IDs: POEM/GPOEM
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Achalasia; Gastroparesis
Keywords: Anesthesia; Pneumoperitoneum; POEM; GPOEM
MeSH Terms: conditions — Esophageal Achalasia; Gastroparesis; Pneumoperitoneum | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: General anesthesia for per-oral endoscopic myotomy — Intra-abdominal pressure measurement

SUMMARY:
The goal of this observational study is to learn about hemodynamic and respiratory repercussions during general anesthesia in patients with achalasia or gastroparesis who underwent an endoscopic treatment such as a peroral endoscopic myotomy (POEM) or gastric (GPOEM).

The main questions it aims to answer are:

* Are there predictable elements reliable to this study-population for the occurrence of adverse events/complications?
* Is there a correlation between the value (percutaneous puncture) of the intra-abdominal pressure and the variations of the patient's respiratory and hemodynamic parameters in the event of a pneumoperitoneum complication?

Participants will be treated with the usual standard of care for this procedure and no additional or specific therapy will be planned for this study.

DETAILED DESCRIPTION:
During the last ten years, the treatment of motor disorders of the esophagus and gastroparesis, by endoscopic approach, has become widespread. Because of its safety and effectiveness, this endoscopic technique has become the gold standard in esophageal and gastric motility disorders. This procedure consists of performing, under general anesthesia, a myotomy of the lower esophageal or pyloric sphincter, by performing a dissection under the mucous membrane beforehand. To properly expose the surgical site, the operator uses CO2, usually at a low flow rate, to reduce the risk of complications. However, subcutaneous emphysema (especially cervical), pneumoperitoneum, pneumothorax and pneumomediastinum occur in about 7.5-55% of cases, according to the literature. These adverse events frequently coincide with anesthetic difficulties. Indeed, the accumulation of CO2 outside the digestive lumen can disrupt mechanical ventilation (restrictive effect) by increasing intra-abdominal or intra-thoracic pressure. Consequently, the inspiratory pressure increases, the tidal volume decreases and the patient can desaturate. Therefore, stopping the endoscopic procedure is necessary and percutaneous CO2 exsufflation is indicated.

The recent evolution of endoscopic treatment improves the future of these patients. However, the anesthetic management during this procedure remains poorly studied and depends mainly on the experience of the responsible physician.

The aims of this prospective study are to be able to explore, on the basis of a detailed analysis of the patient profile (morphological data, medical/surgical history, drug treatment, etc.) and the various aspects of the endoscopic procedure (type of approach, procedure duration, dissection length, etc.), elements predictable for the occurrence of adverse events/complications (pneumoperitoneum, pneumothorax, haemorrhage, etc.); as well as being able to correlate the measurement (percutaneous puncture) of the intra-abdominal pressure to the variations of the respiratory and hemodynamic parameters of the patient in the event of a complication such as pneumoperitoneum. The results of this present project could make it possible to propose a more optimized anesthetic and gastroenterological management protocol for future patients, making it possible to minimize the risk of abdominal distension, as well as its respiratory and hemodynamic consequences.

Potential participants will all be seen, informed and will be offered their participation in the study in preoperative anesthesia consultation, at the Lausanne University Hospital, at least 24 hours before the intervention. Once the eligibility criteria have been verified, the information and consent documents will be presented and detailed. The investigator will explain to each potential participant during the preoperative anesthesia consultation, the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits, and any discomfort it may cause. Each participant will be informed that his/her participation in the study is voluntary and that he/she can withdraw from the study at any time and that the withdrawal of his/her consent will not affect his/her subsequent medical follow-up and treatment. The participant will be informed that his medical file may be examined by authorized persons other than his attending physician. All potential study participants will receive an information sheet and consent form describing the study and providing enough information for the participant to make an informed decision about participating in the study. The patient will have enough time (at least 24 hours) to decide whether or not to participate. If accepted, the consent form will be signed and dated by the investigator or his representative at the same time as the participant's signature on the day of the intervention. A copy of the signed informed consent will be given to the study participant. The consent form will be retained as part of the study records. The anesthetic evaluation during the consultation will always be done according to the criteria in force in our department. At each stage of the study, the patient will have the possibility of contacting an anesthesiologist, in case of questions, and withdrawing their consent to participate in the study without having to justify it.

This study is exploratory in nature, with a primarily descriptive primary objective. The sample size is therefore not based on formal statistical methods. This is rather based on a feasibility estimate of the number of patients that can be included in 24 months by the anesthesiology department. According to the experience of this service, and taking into account the refusal of certain patients to participate in the study, 60 to 150 patients called for endoscopy treatment of the POEM or GPOEM type could be recruited in 24 months. Cases of pneumoperitoneum at the CHUV represent approximately 20% of patients having this type of treatment; we therefore estimate that the data from approximately thirty patients would serve for the exploratory analysis of the secondary objective of correlation between the modifications of the respiratory and hemodynamic parameters and the intra-abdominal pressure values.

The primary objective is to describe the profile of patients in the presence or absence of adverse events. For each of the 2 groups, the following descriptions will be made:

* Continuous variables: minimum, 1st quartile, median, 2nd quartile, maximum (if deemed useful the results will be accompanied by a graphic representation: box-plot, dot-plot or violin plot)
* Qualitative variable: frequency and proportion per group

The secondary objectives are:

1. Identify predictors of adverse events/complications

   A logistic regression will be performed using a regularization method (lasso, elastic net) or by selecting a restricted set of variables (3 maximum). As this analysis is exploratory, and therefore, before fitting any type of regression model, the primary analysis described above will help to understand which models can be fitted, which covariate might or might not be included in the model.
2. Correlate changes in respiratory and hemodynamic parameters to intra-abdominal pressure values

The factors studied will be the respiratory parameters (ventilatory mode, peak pressure, plateau pressure, tidal volume, pressure support level, respiratory rate, PEEP, FiO2, SpO2 and exhaled CO2) and hemodynamic values (mean arterial pressure, heart rate and use of vasopressors) throughout the endoscopic procedure. Correlations will be made on the subgroup of patients who have had pneumoperitoneum (estimate of about thirty patients). The Pearson and Spearman correlation coefficients as well as their 95% confidence intervals will be provided for the correlations between the continuous variables, the qualitative ones, respectively. For correlations between continuous and qualitative variables, the logistic regression method will be applied. The contingency tables will be presented in the case of two qualitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Completed and signed consent form (consent form attached)
* Age ≥ 18 years old
* Anesthetic risk classification according to ASA, from 1 to 3
* Patients summoned for POEM or GPOEM type endoscopy treatment

Exclusion Criteria:

- Inability to follow study procedures, eg. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with achalasia or gastroparesis who are summoned for POEM or GPOEM type endoscopy treatment at the Lausanne University Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Describe in detail the profile of operated patients and the various characteristics of the endoscopic procedure, in the presence or absence of adverse events/complications. | 48 hours

SECONDARY OUTCOMES:
Verify the presence of predictable elements of adverse events | 48 hours
Look for a correlation between the modifications of the respiratory and hemodynamic parameters with the values of intra-abdominal pressure measured, during the exsufflations by stages of the pneumoperitoneums | 48hours

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Chollet-Rivier, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bang YS, Park C. Anesthetic Consideration for Peroral Endoscopic Myotomy. Clin Endosc. 2019 Nov;52(6):549-555. doi: 10.5946/ce.2019.033. Epub 2019 Jul 10. PMID 31288505
- [Result] Darisetty S, Nabi Z, Ramchandani M, Chavan R, Kotla R, Nageshwar Reddy D. Anesthesia in per-oral endoscopic myotomy: A large tertiary care centre experience. Indian J Gastroenterol. 2017 Jul;36(4):305-312. doi: 10.1007/s12664-017-0782-0. Epub 2017 Aug 24. PMID 28840505
- [Result] Jayan N, Jacob JS, Mathew M, Mukkada RJ. Anesthesia for peroral endoscopic myotomy: A retrospective case series. J Anaesthesiol Clin Pharmacol. 2016 Jul-Sep;32(3):379-81. doi: 10.4103/0970-9185.188829. PMID 27625490
- [Result] Loser B, Werner YB, Punke MA, Saugel B, Haas S, Reuter DA, Mann O, Dupree A, Schachschal G, Rosch T, Petzoldt M. Anesthetic considerations for patients with esophageal achalasia undergoing peroral endoscopic myotomy: a retrospective case series review. Can J Anaesth. 2017 May;64(5):480-488. doi: 10.1007/s12630-017-0820-5. Epub 2017 Jan 23. PMID 28116675
- [Result] Nishihara Y, Yoshida T, Ooi M, Obata N, Izuta S, Mizobuchi S. Anesthetic management and associated complications of peroral endoscopic myotomy: A case series. World J Gastrointest Endosc. 2018 Sep 16;10(9):193-199. doi: 10.4253/wjge.v10.i9.193. PMID 30283602
- [Result] Okada T, Izuta S, Mizobuchi S. A case of ventilatory impairment during per-oral endoscopic myotomy under general anesthesia. JA Clin Rep. 2018 Feb 26;4(1):23. doi: 10.1186/s40981-018-0160-7. PMID 32026954
- [Result] Podboy A, Hwang JH, Nguyen LA, Garcia P, Zikos TA, Kamal A, Triadafilopoulos G, Clarke JO. Gastric per-oral endoscopic myotomy: Current status and future directions. World J Gastroenterol. 2019 Jun 7;25(21):2581-2590. doi: 10.3748/wjg.v25.i21.2581. PMID 31210711
- [Result] Sosa G, Gandham N, Landeras V, Calimag AP, Lerma E. Abdominal compartment syndrome. Dis Mon. 2019 Jan;65(1):5-19. doi: 10.1016/j.disamonth.2018.04.003. Epub 2018 Nov 17. No abstract available. PMID 30454823
- [Result] Werner YB, von Renteln D, Noder T, Schachschal G, Denzer UW, Groth S, Nast JF, Kersten JF, Petzoldt M, Adam G, Mann O, Repici A, Hassan C, Rosch T. Early adverse events of per-oral endoscopic myotomy. Gastrointest Endosc. 2017 Apr;85(4):708-718.e2. doi: 10.1016/j.gie.2016.08.033. Epub 2016 Sep 5. PMID 27609778
- [Result] Maunder RJ, Pierson DJ, Hudson LD. Subcutaneous and mediastinal emphysema. Pathophysiology, diagnosis, and management. Arch Intern Med. 1984 Jul;144(7):1447-53. PMID 6375617